CLINICAL TRIAL: NCT06353074
Title: Uterine Preservation With Acar's Atony Suture for Postpartum Uterine Atony
Brief Title: Uterine Preservation With Acar's Atony Suture for Postpartum Uterine Hemorrhage
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Cemre Alan, Fellow of Gynecologic Oncology, Necmettin Erbakan University
Other Study IDs: 1335cemre.
Record Dates: First submitted 2023-12-26; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Uterine Atony With Hemorrhage; Postpartum Hemorrhage
Keywords: Cesarean section; compression suture; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: The patients who had uterine atony during delivery and to whom Acar's atony suture were performed consisted study group.

SUMMARY:
This study is aimed to show effectiveness of a new suture technique to stop postpartum uterine bleeding due to uterine atony.

DETAILED DESCRIPTION:
A retrospective study of all women received Acar's uterine compressive atony suture between January 2021-November 2023 at a single tertiary hospital with approximately 4000 deliveries per year, was performed. The local protocol for PPH due to uterine atony is uterine manual compression, 20 IU of intravenous oxytocin in 500 cc of normal saline at 500 cc/h; 800 µg of misoprostol inserted per rectal. If additional treatment is needed, carbetocin 100mcg in 100 cc of normal saline or tranexamic acid in different posologies are used.

If uterine atony persists, intrauterine balloon tamponade or uterine compressive sutures were applied at the discretion of the physician and according to mode of delivery. When uterine compressive suture was performed, original Acar's atony suture was applied.

ELIGIBILITY:
Inclusion Criteria:

* women without systemic disease

Exclusion Criteria:

* cardiac disease
* rheumatological disease

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women admitted to the university hospital for delivery and women referred to the university hospital with uterine atony diagnosis
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Postpartum hysterectomy and/or intensive care unit need ratio | Since first operation to discharge from hospital assessed up to 5 days
  The need for hysterectomy or massive transfusion because of unstoppable and mortal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ali Acar, Clinic Prof., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Cemre Alan, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. Because the investigators want to see long term results first and larger sample sizes.

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Santos RR, Martins I, Clode N, Santo S. Uterine preservation with Alcides-Pereira's compressive sutures for postpartum uterine atony. Eur J Obstet Gynecol Reprod Biol. 2022 Oct;277:27-31. doi: 10.1016/j.ejogrb.2022.08.008. Epub 2022 Aug 12. PMID 35987075
- [Background] Balki M, Wong CA. Refractory uterine atony: still a problem after all these years. Int J Obstet Anesth. 2021 Nov;48:103207. doi: 10.1016/j.ijoa.2021.103207. Epub 2021 Jul 21. PMID 34391025
- [Background] Bateman BT, Berman MF, Riley LE, Leffert LR. The epidemiology of postpartum hemorrhage in a large, nationwide sample of deliveries. Anesth Analg. 2010 May 1;110(5):1368-73. doi: 10.1213/ANE.0b013e3181d74898. Epub 2010 Mar 17. PMID 20237047
- [Background] Al-Zirqi I, Vangen S, Forsen L, Stray-Pedersen B. Prevalence and risk factors of severe obstetric haemorrhage. BJOG. 2008 Sep;115(10):1265-72. doi: 10.1111/j.1471-0528.2008.01859.x. PMID 18715412
- [Background] Ramler PI, van den Akker T, Henriquez DDCA, Zwart JJ, van Roosmalen J, van Lith JMM, van der Bom JG; TeMpOH-1 study group. Women receiving massive transfusion due to postpartum hemorrhage: A comparison over time between two nationwide cohort studies. Acta Obstet Gynecol Scand. 2019 Jun;98(6):795-804. doi: 10.1111/aogs.13542. Epub 2019 Feb 11. PMID 30667050
- [Background] Huque S, Roberts I, Fawole B, Chaudhri R, Arulkumaran S, Shakur-Still H. Risk factors for peripartum hysterectomy among women with postpartum haemorrhage: analysis of data from the WOMAN trial. BMC Pregnancy Childbirth. 2018 May 29;18(1):186. doi: 10.1186/s12884-018-1829-7. PMID 29843627
- [Background] B-Lynch C, Coker A, Lawal AH, Abu J, Cowen MJ. The B-Lynch surgical technique for the control of massive postpartum haemorrhage: an alternative to hysterectomy? Five cases reported. Br J Obstet Gynaecol. 1997 Mar;104(3):372-5. doi: 10.1111/j.1471-0528.1997.tb11471.x. PMID 9091019
- [Background] Nelson WL, O'Brien JM. The uterine sandwich for persistent uterine atony: combining the B-Lynch compression suture and an intrauterine Bakri balloon. Am J Obstet Gynecol. 2007 May;196(5):e9-10. doi: 10.1016/j.ajog.2006.10.887. PMID 17466689
- [Background] Baskett TF. Uterine compression sutures for postpartum hemorrhage: efficacy, morbidity, and subsequent pregnancy. Obstet Gynecol. 2007 Jul;110(1):68-71. doi: 10.1097/01.AOG.0000267499.40531.a4. PMID 17601898
- [Background] Acar A, Ercan F, Pekin A, Elci Atilgan A, Sayal HB, Balci O, Gorkemli H. Conservative management of placental invasion anomalies with an intracavitary suture technique. Int J Gynaecol Obstet. 2018 Nov;143(2):184-190. doi: 10.1002/ijgo.12593. Epub 2018 Aug 13. PMID 29989156
- [Background] Pereira A, Nunes F, Pedroso S, Saraiva J, Retto H, Meirinho M. Compressive uterine sutures to treat postpartum bleeding secondary to uterine atony. Obstet Gynecol. 2005 Sep;106(3):569-72. doi: 10.1097/01.AOG.0000168434.28222.d3. PMID 16135589
- [Background] Moleiro ML, Braga J, Machado MJ, Guedes-Martins L. Uterine Compression Sutures in Controlling Postpartum Haemorrhage: A Narrative Review. Acta Med Port. 2022 Jan 3;35(1):51-58. doi: 10.20344/amp.11987. Epub 2019 Oct 7. PMID 32208130
- [Derived] Acar A, Alan C, Dogru S. A new technique: Acar's atony suture for postpartum uterine hemorrhage. Z Geburtshilfe Neonatol. 2025 Jun;229(3):195-200. doi: 10.1055/a-2441-6846. Epub 2024 Nov 11. PMID 39529317